CLINICAL TRIAL: NCT02496676
Title: A Double-blind, Placebo-controlled, Crossover Study of Magnesium Supplementation in Patients With XMEN Syndrome
Brief Title: Magnesium Supplementation in People With XMEN Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 150161; 15-I-0161 (Other: National Institutes of Health)
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Results first posted 2022-01-26 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2020-04

CONDITIONS: XMEN
Keywords: Neoplasia; magnesium transporter 1 (MAGT1); Primary Immunodeficiency; X-linked immunodeficiency; Epstein-Barr virus (EBV) infection
MeSH Terms: conditions — Neoplasms; Primary Immunodeficiency Diseases; Epstein-Barr Virus Infections; Infections | interventions — threonic acid; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Magnesium, then placebo (Active Comparator): In phase 1, participants received oral magnesium L-threonate for 12 weeks then crossover to placebo for 12 weeks, followed by a 2-week washout period. In phase 2, all participants received 3 days of intravenous MgSO4 in 3 daily doses totaling 30 mg/kg/day followed by oral magnesium L-threonate for 24 weeks.
  Interventions: Dietary Supplement: Magnesium L-threonate; Other: Placebo; Drug: Intravenous (IV) magnesium sulfate (MgSO4)
- Placebo, then magnesium (Placebo Comparator): In phase 1, participants received oral placebo for 12 weeks then crossover to oral magnesium L-threonate for 12 weeks, followed by a 2-week washout period. In phase 2, all participants received 3 days of intravenous MgSO4 in 3 daily doses totaling 30 mg/kg/day followed by oral magnesium L-threonate for 24 weeks.
  Interventions: Dietary Supplement: Magnesium L-threonate; Other: Placebo; Drug: Intravenous (IV) magnesium sulfate (MgSO4)

INTERVENTIONS:
Dietary Supplement: Magnesium L-threonate — In Part I, participants will receive 12 weeks of oral magnesium L-threonate; will be dose escalated based on weight.
  In Part 2, participants will receive 24 weeks of oral magnesium L-threonate; will be dose escalated based on weight.
Other: Placebo — In Part I, participants will receive 12 weeks of oral placebo; will be dose escalated based on weight.
Drug: Intravenous (IV) magnesium sulfate (MgSO4) — In Part II, participants will be hospitalized to receive 3 days of IV magnesium sulfate (MgS04).

SUMMARY:
Background:

- X-linked immunodeficiency with magnesium defect, Epstein-Barr virus infection, and neoplasia syndrome is called XMEN syndrome. In this genetic condition, the cells have less magnesium than normal. This makes it hard for the body to fight infections. Researchers want to see if magnesium supplements can make it easier for the body to fight infection.

Objective:

- To see if magnesium supplements can strengthen the immune system and reduce the amount of Epstein-Barr virus in people with XMEN syndrome.

Eligibility:

- People ages 6 and older who have XMEN syndrome

Design:

* Participants will be screened with:
* Medical history
* Physical exam
* CT scan: Participants will drink a contrast and may get dye through an IV in the arm. They will lie in a machine that takes pictures of the body.
* EKG: Small sticky patches on the body will trace heart rhythm.
* Blood tests
* The study has 2 parts.
* Participants doing both parts will participate for 1 year and visit the clinic about 15 times. These visits will include a physical exam and blood and urine tests.
* Participants doing only the first part finish in 6 months and have fewer visits.
* For study part 1, participants will take magnesium pills for 3 months and placebo pills for another 3 months.
* At 3 and 6 months, they will have physical exam, medical history, blood and urine tests, and an EKG.
* If the magnesium pills are not helpful, participants will do study part 2.
* They will be admitted to the hospital for 4 5 days to get magnesium for 3 days through an arm vein.
* They will take magnesium pills for another 6 months.

DETAILED DESCRIPTION:
X-linked immunodeficiency magnesium defect, Epstein-Barr virus (EBV) infection and neoplasia (XMEN) syndrome is a primary immunodeficiency caused by the loss of expression of the magnesium transporter 1 (MAGT1). This syndrome is associated with cluster of differentiation 4 (CD4) lymphopenia, chronic EBV infection in most patients, and EBV-related lymphoproliferative disorders. The loss of MAGT1 leads to impaired T cell activation and decreased expression of the activator receptor, NKG2D on natural killer (NK) cells and CD8 T cells, leading to decreased EBV-specific cytolytic function of these cells. Results of previous studies suggest that magnesium supplementation may be a viable therapeutic option for patients with XMEN.

The proposed study has 2 parts, and patients will be divided into 2 cohorts. Patients in cohort 1 (high EBV group) will have baseline blood EBV viral load greater than or equal to 5,000 copies/mL or EBV log greater than or equal to 3.7 IU/mL. Patients in cohort 2 (low/no EBV group) will have baseline blood EBV viral load <5,000 copies/mL or EBV log <3.7 IU/mL. Part I is a randomized, double-blind, placebo-controlled, crossover study to evaluate the safety and efficacy of oral magnesium L-threonate in patients with XMEN syndrome. Within each cohort, patients will be randomized to receive escalating doses of either placebo or oral magnesium L-threonate for 12 weeks. Patients will then receive the crossover treatment (magnesium or placebo) for an additional 12 weeks. For patients who experience a 0.5-log decrease in the number of EBV-infected B cells (cohort 1) or a greater than or equal to 2-fold increase in NKG2D receptor expression on cluster of differentiation 8 (CD8+) T cells (cohort 2) with oral magnesium as compared to placebo, the study will be complete. Patients who do not meet this efficacy outcome will undergo a 2-week washout period and proceed to Part II, an open-label, non-randomized evaluation of intravenous magnesium sulfate (MgSO4) followed by oral magnesium L-threonate. These patients will be hospitalized to receive 3 days of intravenous MgSO4 in 3 daily doses totaling 30 mg/kg/day. They will then restart escalating doses of oral magnesium L-threonate and continue for the remaining 24 weeks of Part II. If conducted, Part II will allow for secondary analyses to compare different durations of magnesium supplementation.

ELIGIBILITY:
* INCLUSION CRITERIA:

All of the following inclusion criteria must be met prior to enrollment:

1. Molecular diagnosis of the MAGT1 genetic defect
2. Greater than or equal to 6 years years of age
3. Willingness to stop magnesium supplements (other than the study agent) and any multivitamins or over-the counter-supplements that may contain magnesium for the duration of the study
4. Willingness to go without magnesium supplementation during a 12-week placebo period and during both 2-week washout periods (pre-study and mid-study)
5. Willingness to have samples stored for future research
6. Must have a physician at home for follow-up care

EXCLUSION CRITERIA:

1. Chemotherapy or radiotherapy for lymphoma within 12 months prior to enrollment
2. Rituximab exposure within 6 months prior to enrollment
3. Systemic symptoms suggestive of evolving lymphoma
4. History of clinically significant cardiac arrhythmias or cardiac defects
5. Renal insufficiency (calculated creatinine clearance <50 mL/min or insufficiency requiring dialysis)
6. Advanced heart block
7. Hypermagnesemia, defined as magnesium serum concentrations >2 mmol/L (>5 mg/dL)
8. Human immunodeficiency virus (HIV) seropositivity
9. Signs or symptoms of life-threatening active microbial infection
10. History of hypersensitivity to any of the study agents
11. Any condition that, in the investigator s opinion, may substantially increase the risk associated with study participation or compromise the study s scientific objectives
12. Participation in a clinical protocol which includes an intervention that, in the opinion of the investigator, may affect the results of the current study

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Ravell Aumaitre, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Li FY, Chaigne-Delalande B, Kanellopoulou C, Davis JC, Matthews HF, Douek DC, Cohen JI, Uzel G, Su HC, Lenardo MJ. Second messenger role for Mg2+ revealed by human T-cell immunodeficiency. Nature. 2011 Jul 27;475(7357):471-6. doi: 10.1038/nature10246. PMID 21796205
- [Background] Chaigne-Delalande B, Li FY, O'Connor GM, Lukacs MJ, Jiang P, Zheng L, Shatzer A, Biancalana M, Pittaluga S, Matthews HF, Jancel TJ, Bleesing JJ, Marsh RA, Kuijpers TW, Nichols KE, Lucas CL, Nagpal S, Mehmet H, Su HC, Cohen JI, Uzel G, Lenardo MJ. Mg2+ regulates cytotoxic functions of NK and CD8 T cells in chronic EBV infection through NKG2D. Science. 2013 Jul 12;341(6142):186-91. doi: 10.1126/science.1240094. PMID 23846901
- [Background] Li FY, Chaigne-Delalande B, Su H, Uzel G, Matthews H, Lenardo MJ. XMEN disease: a new primary immunodeficiency affecting Mg2+ regulation of immunity against Epstein-Barr virus. Blood. 2014 Apr 3;123(14):2148-52. doi: 10.1182/blood-2013-11-538686. Epub 2014 Feb 18. PMID 24550228
- [Result] Chauvin SD, Price S, Zou J, Hunsberger S, Brofferio A, Matthews H, Similuk M, Rosenzweig SD, Su HC, Cohen JI, Lenardo MJ, Ravell JC. A Double-Blind, Placebo-Controlled, Crossover Study of Magnesium Supplementation in Patients with XMEN Disease. J Clin Immunol. 2022 Jan;42(1):108-118. doi: 10.1007/s10875-021-01137-w. Epub 2021 Oct 16. PMID 34655400
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-I-0161.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8 participants were consented to protocol. 2 participants did not meet inclusion criteria and one participant declined to participate.
Period: Phase 1 - Period 1
Arm/Group | Magnesium, Then Placebo | Placebo, Then Magnesium
Started | 2 | 3
Completed | 2 | 2
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Phase 1 - Period 2
Arm/Group | Magnesium, Then Placebo | Placebo, Then Magnesium
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Magnesium, Then Placebo | Placebo, Then Magnesium
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Phase 2 - IV MgSO4
Arm/Group | Magnesium, Then Placebo | Placebo, Then Magnesium
Started | 2 | 2
Completed | 2 | 1
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Phase 2 - Oral Magnesium
Arm/Group | Magnesium, Then Placebo | Placebo, Then Magnesium
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium, Then Placebo | Placebo, Then Magnesium | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Participants With a ≥0.5 Log Reduction in the Number of EBV-infected B Cells After Magnesium Supplementation as Compared to Placebo - Phase 1
Description: Participants with a ≥ 0.5 log decrease in the absolute number of Epstein-Barr virus (EBV) infected B-cells by flow cytometric Fluorescence in situ hybridization (FISH) assay after 12 weeks of oral magnesium supplementation compared to 12 weeks of placebo.
Time Frame: After 12 weeks of each intervention
Population: The analyses included only EBV positive subject who completed Phase 1 of the study. In this phase, two participants were EBV positive, but only one participant completed Phase 1.
Measure: Count of Participants; unit: Participants
Groups:
- Magnesium: Participants received oral magnesium L-threonate for 12 weeks
- Placebo: Participants received oral placebo for 12 weeks
Arm/Group | Magnesium | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

2. Primary Outcome: Participants With 2-fold or Greater Increase in NKG2D Expression in CD8 T+ Cells After Magnesium Supplementation as Compared to Placebo - Phase 1
Description: Participants with difference of a 2-fold or greater increase in NKG2D expression in cluster of differentiation 8 (CD8+) T cells after 12 weeks of oral magnesium supplementation versus 12 weeks of placebo.
Time Frame: After 12 weeks of each intervention
Population: The analyses included only EBV negative subjects who completed phase 1 of the study, which is the crossover phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Magnesium | Placebo
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

3. Secondary Outcome: Participants With 2-fold or Greater Increase in NKG2D Expression in CD8 T+ Cells After Magnesium Supplementation as Compared to Placebo - Phase 1
Description: as for outcome 2
Time Frame: After 12 weeks of each intervention
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Magnesium | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

4. Secondary Outcome: Participants With a Decrease in the Absolute Number of EBV Infected B Cells Before and After Magnesium Supplementation - Phase 2
Description: Participants with a ≥ 0.5 log decrease in the absolute number of Epstein-Barr virus (EBV) infected B-cells by flow cytometric Fluorescence in situ hybridization (FISH) assay before and after 24 weeks of magnesium supplementation
Time Frame: 24 weeks, during phase 2 of study
Population: Analysis included all EBV positive participants who completed phase 2 of study
Measure: Count of Participants; unit: Participants
Groups:
- Magnesium: In phase 2, participants received 3 days of intravenous MgSO4 daily at 30 mg/kg/day followed by oral magnesium L-threonate for 24 weeks.
Arm/Group | Magnesium
Number analyzed (Participants) | 1
Participants | 0

5. Secondary Outcome: Participants With 2-fold or Greater Increase in NKG2D Expression in CD8 T+ Cells Before and After Magnesium Supplementation - Phase 2
Description: Participants with a 2-fold or greater increase in NKG2D expression in CD8+ T cells before and after magnesium supplementation for 24 weeks in phase 2 of study
Time Frame: 24 weeks, during phase 2 of study
Population: Analysis included all participants who completed phase 2 of study
Measure: Count of Participants; unit: Participants
Arm/Group | Magnesium
Number analyzed (Participants) | 3
Participants | 0

6. Secondary Outcome: Participants With Adverse Events by Grade
Description: Participants with adverse events by grade using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE, version 4) grading criteria.
  * Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; no intervention indicated
  * Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL)
  * Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL
  * Grade 4 Life-threatening consequences; urgent intervention indicated
  * Grade 5 Death related to adverse event (AE)
Time Frame: 1 year
Population: Analysis included all subjects who started each arm of the study
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 - Oral Magnesium: In phase 1, participants received oral magnesium L-threonate for 12 weeks
- Phase 1 - Placebo: Participants received oral placebo for 12 weeks
- Phase 2 - IV MgSO4: In phase 2, participants received 3 days of intravenous MgSO4 in 3 daily doses totaling 30 mg/kg/day
- Phase 2 - Oral Magnesium: In phase 2, participants received oral magnesium L-threonate for 24 weeks.
Arm/Group | Phase 1 - Oral Magnesium | Phase 1 - Placebo | Phase 2 - IV MgSO4 | Phase 2 - Oral Magnesium
Number analyzed (Participants) | 4 | 5 | 4 | 3
Participants
  Grade 1 | 4 | 4 | 1 | 2
  Grade 2 | 1 | 3 | 1 | 3
  Grade 3 | 0 | 2 | 1 | 0
  Grade 4 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0

7. Secondary Outcome: Participants With Severe Adverse Events
Description: Participants with severe adverse events using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE, version 4) to evaluate severity.
Time Frame: 1 year
Population: Analysis included all subjects who started each arm of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - Oral Magnesium | Phase 1 - Placebo | Phase 2 - IV MgSO4 | Phase 2 - Oral Magnesium
Number analyzed (Participants) | 4 | 5 | 4 | 3
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Phase 1 - Oral Magnesium | Phase 1 - Placebo | Phase 2 - IV MgSO4 | Phase 2 - Oral Magnesium
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 1/4 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 - Oral Magnesium (N=4) | Phase 1 - Placebo (N=5) | Phase 2 - IV MgSO4 (N=4) | Phase 2 - Oral Magnesium (N=3)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 3 (8) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (13) | 3 (14) | 0 (0) | 1 (2)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT02496676/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT02496676/ICF_001.pdf